CLINICAL TRIAL: NCT01789047
Title: Topiramate as an Adjunct to Amantadine in the Treatment of Dyskinesia in Parkinson's Disease
Acronym: TOP-DYSK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: Rush University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Christopher G. Goetz, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP-DYSK
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Idiopathic Parkinson's Disease; Drug Induced Dyskinesia
Keywords: Parkinson's disease; dyskinesia; Indonesia; amantadine
MeSH Terms: conditions — Parkinson Disease; Dyskinesia, Drug-Induced; Dyskinesias | interventions — Topiramate; Sugars; Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Active Comparator): Topiramate as adjunct to amantadine.
  Interventions: Drug: Topiramate; Drug: Amantadine
- Placebo (sugar pill) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Drug: Amantadine

INTERVENTIONS:
Drug: Topiramate — Topiramate as adjunct to amantadine
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — Placebo control
  Other Names: sugar pill
  Arms: Placebo (sugar pill)
Drug: Amantadine — Existing treatment for all participants
  Other Names: Symmetrel

SUMMARY:
The study will involve an eighteen-week, double-blind, placebo-controlled parallel designed comparison between add-on topiramate and add-on placebo to stable treatment with amatadine in the treatment of Parkinson's disease (PD) patients who continue to have dyskinesia on amantadine.

DETAILED DESCRIPTION:
We conducted a randomized placebo controlled trial of topiramate in PD dyskinetic subjects already on amantadine but with continuing dyskinesia. Topiramate or placebo was introduced in blinded fashion with a gradual titration (topiramate 25-150 mg/d) over 6 weeks and then a maintenance period of 8 weeks. The primary outcome of interest was change from baseline to end of study in total Unified Dyskinesia Rating Scale (UDysRS) score using Intention to Treat analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease patient, defined by United Kingdom (UK) Brain Bank criteria
2. Current age between 30-90
3. Clinically pertinent dyskinesias defined by Clinical Global Impression - Severity (CGI-s) score (see attachment) > 3 (mild) established by clinician's total assessment of patient including objective observation during the screening process. *
4. Stable doses of all antiparkinsonian medications for at least 4 weeks
5. Stable treatment with at least 200 mg amantadine for at least 4 weeks.
6. Presence of a caregiver willing to participate in the study
7. In the opinion of the enrolling investigator, the subject will be able to maintain current dosing schedule of antiparkinsonian drugs for the duration of the trial.
8. Subjects must be free of dementia, depression and psychosis as determined by clinical examination.
9. The subject must be willing to participate in all study related activities and visits.

Exclusion criteria:

1. Any subjects with clinical evidence suggestive of an atypical or secondary form of Parkinson's Disease
2. Any subject who, in the opinion of the Principal Investigator, has a concomitant medical illness which would preclude them from being treated with amantadine,
3. Any subject who, in the opinion of the Principal Investigator, will be unable to maintain current stable dosing of their anti-parkinsonian medications for the duration of the trial,
4. Any subject with evidence for dementia, depression, or psychosis, as determined by clinical examination.
5. Any subject who has not signed informed consent, or unable or unwilling to participate in all of the study related activities.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Goetz, MD, Principal Investigator — Rush University Medical Center
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Placebo (Sugar Pill)
Started | 21 | 21
Completed | 17 | 17
Not Completed | 4 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (6.9) | 63.1 (8.9) | 62.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 15 | 12 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: The Unified Dyskinesia Rating Scale (UDysRS)
Description: The Unified Dyskinesia Rating Scale (UDysRS) will be the primary outcome measure for this study. This choice is based on the outcome of the Validation of Dyskinesia Rating Scales study. In this study, the UDysRS was identified as the most sensitive scale to detect change in dyskinesia in an 8-week, double-blind, placebo-controlled trial of amatadine. The UDysRS utilizes rater information, patient self-report and objective measures of dyskinesia to provide assessments of impairment and disability due to dyskinesia. Score ranges are 0-108 with higher scores representing more severe impairment.
Time Frame: Change from baseline to week 14 (end of study) on the Unified Dyskinesia Rating Scale
Population: Last Observation Carried Forward imputation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate | Placebo (Sugar Pill)
Number analyzed (Participants) | 21 | 21
units on a scale | 4.00 (11.34) | 1.67 (10.27)

2. Other Pre Specified Outcome: Clinical Global Impression - Change Score
Description: The Clinical Global Impression - Change score is an ordinal measure of change with a range of 0 (not assessed) to 7 (very much worse). A score of 4 is associated with "no change".
Time Frame: Assessed at Week 10 and 14 by blinded treating physician and subject
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: This is a 4-part scale that rates both non-motor and motor (including dyskinesia) aspects of Parkinson's disease. Parts of the scales will be completed by the blinded treating physician while assessing the subject and other parts will be self-completed by the subject
Time Frame: Assessed at baseline, week 6, week 10 and week 14
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Hoehn & Yahr Staging
Description: Hoehn & Yahr staging of Parkinson's disease is completed by the blinded treating physician assessing the subject
Time Frame: Assessment completed at baseline, week 6, week 10 and week 14
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Topiramate | Placebo (Sugar Pill)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/21
Other Adverse Events (participants affected / at risk) | 16/21 | 12/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=21) | Placebo (Sugar Pill) (N=21)
Transit Ischemic Attack-like symptoms (Nervous system disorders) | 1 (1) | 0 (0) — Recovered without treatment
Fall leading to hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Recovered with treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=21) | Placebo (Sugar Pill) (N=21)
Balance instability (Nervous system disorders) | 1 (1) | 1 (1)
Biting lower lip (General disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 3 (3) | 1 (1)
cognitive decline (Nervous system disorders) | 0 (0) | 1 (1)
Common cold (Infections and infestations) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 2 (2)
Falls (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2) | 2 (2)
Headache (General disorders) | 1 (1) | 0 (0)
Increased OFF time (Nervous system disorders) | 2 (2) | 3 (3)
Increased dreaming (Nervous system disorders) | 0 (0) | 1 (1)
Increased freezing of gait (Nervous system disorders) | 0 (0) | 1 (1)
Intermittent SOB (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ottis media (Infections and infestations) | 1 (1) | 0 (0)
Pre cancerous lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 2 (2)
Speech abnormalities (Nervous system disorders) | 1 (1) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Tingling fingers and toes (General disorders) | 1 (1) | 0 (0)
Worsening constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No